CLINICAL TRIAL: NCT00920465
Title: Comparison of the Effectiveness of Abortive Measures From the Administration of Mifegyne and Cytotec at One and Two Visits
Brief Title: Treatment Regimens for Mifegyne and Cytotec
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Western Galilee Hospital-Nahariya (Other Government)
Responsible Party: Dr. Renee Tendler, Western Galilee Hospital-Nahariya
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 4-10-2007
Record Dates: First submitted 2009-06-12; First posted 2009-06-15 (Estimated); Last update posted 2011-05-25 (Estimated); Status verified 2010-11

CONDITIONS: Medical Abortion
MeSH Terms: interventions — Mifepristone; Misoprostol

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- one-visit (Experimental)
  Interventions: Drug: mifegyne and cytotec
- two-visit (Active Comparator)
  Interventions: Drug: mifegyne and cytotec

INTERVENTIONS:
Drug: mifegyne and cytotec — One day dosage versus two days dosage
  Other Names: Comparison of one day dosing to two days dosing

SUMMARY:
The purpose of this study is to test two regimens of mifegyne and cytotec for medical abortion. The investigators hypothesize that administration of both medications during one hospital visit will not compromise effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* above age 18,
* for whom Mifegyne and cytotec are indicated.

Exclusion Criteria:

* inflammation of oral cavity.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2009-06; Primary Completion 2011-12 (Estimated); Study Completion 2011-12 (Estimated)

PRIMARY OUTCOMES:
percentage of complete abortion | one month

CONTACTS AND LOCATIONS:
Locations (1):
- Western Galilee Hospital- Nahariya, Nahariya, Israel